CLINICAL TRIAL: NCT05260541
Title: A Phase 2, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of PRAX-114 in Participants With Post-Traumatic Stress Disorder
Brief Title: A Clinical Trial of PRAX-114 in Participants With Post-Traumatic Stress Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer developing for this indication
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-114-221
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Post-traumatic Stress Disorder; Post Traumatic Stress Disorder; Stress Disorder; Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Mental Disorder
Keywords: Agents, GABA; Receptors, GABA-A; Allosteric Regulation; PRAX-114
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blind PRAX-114 (Experimental): Double-blind period - 40 or 60 mg PRAX-114 once daily in the evening
  Interventions: Drug: 60 mg PRAX-114 or 40 mg PRAX-114
- Double-blind Placebo (Placebo Comparator): Double-blind period - placebo once daily in the evening
  Interventions: Drug: Placebo
- Open-label Extension PRAX-114 (Experimental): Open-label extension period - 40 mg PRAX-114 once daily in the evening
  Interventions: Drug: 40 mg PRAX-114

INTERVENTIONS:
Drug: 60 mg PRAX-114 or 40 mg PRAX-114 — Once daily oral treatment for 4 weeks
  Arms: Double-blind PRAX-114
Drug: Placebo — Once daily oral treatment for 4 weeks
  Arms: Double-blind Placebo
Drug: 40 mg PRAX-114 — Once daily oral treatment for 8 weeks
  Arms: Open-label Extension PRAX-114

SUMMARY:
This trial is comprised of a 4-week randomized, double-blind, placebo-controlled treatment period followed by an optional 8-week open-label extension (OLE) period.

This trial will evaluate the efficacy and safety of oral PRAX-114 flexibly dosed at 40 to 60 mg for 4 weeks compared to placebo in adults with PTSD. The OLE period consisting of treatment with 40 mg PRAX-114 for 8 weeks will provide additional efficacy and safety data.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of PTSD with duration >6 months, as confirmed by psychiatric evaluation.
2. CAPS-5 total score ≥30 at Screening and Baseline.
3. Body mass index (BMI) of 18 to 38 kg/m2.

Exclusion Criteria:

1. Experienced the index traumatic event before age 16.
2. Has an active legal, worker's compensation, or disability claim for PTSD.
3. Lifetime history of bipolar disorder, a psychotic disorder (eg, schizophrenia or schizoaffective disorder), or obsessive-compulsive disorder or a history of a psychotic mood episode in last 2 years.
4. HAM-D17 score of >18 at Screening or Baseline.
5. Any current psychiatric disorder (other than PTSD).
6. Lifetime history of seizures, including febrile seizures.
7. Daily consumption of more than 2 standard alcohol-containing beverages for males or more than 1 standard alcohol-containing beverages for females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total score at Day 29 | 29 days
  The CAPS-5 is a clinician-rated PTSD rating scale consisting of 30 items; the total score is calculated as the sum of 20 items assessing the 20 DSM-5 PTSD symptoms. These symptom items are scored on a 5-point scale from 0 (absent) to 4 (extreme/incapacitating). The total score of the 20 items ranges from 0 to 80 with higher scores indicating more severe PTSD symptoms. Therefore, a decrease in the total score indicates symptom improvement.

SECONDARY OUTCOMES:
Change from baseline in the CAPS-5 total score at Day 15 and 43 | 15 days and 43 days
  The CAPS-5 is a clinician-rated PTSD rating scale consisting of 30 items; the total score is calculated as the sum of 20 items assessing the 20 DSM-5 PTSD symptoms. These symptom items are scored on a 5-point scale from 0 (absent) to 4 (extreme/incapacitating). The total score of the 20 items ranges from 0 to 80 with higher scores indicating more severe PTSD symptoms. Therefore, a decrease in the total score indicates symptom improvement.
Change from baseline in Clinical Global Impression-Severity (CGI-S) score at Day 29, Day 15, and Day 43 | 15 days, 29 days, and 43 days
  The CGI-S assesses the clinician's impression of the participant's current depression symptoms. The clinician should use his/her total clinical experience with this patient population and rate the current severity of the participant's mental illness on a 7-point scale from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients).
Change from baseline in Clinical Global Impression-Improvement (CGI-I) score at Day 29, Day 15, and Day 43 | 15 days, 29 days, and 43 days
  The CGI-I assesses the participant's improvement (or worsening). The clinician is required to assess the participant's condition relative to Baseline (Day 1) on a 7-point scale from 1 (Very much improved) to 7 (Very much worse).
Change from baseline in the CAPS-5 symptom cluster scores at Day 29, Day 15, and Day 43 | 15 days, 29 days, and 43 days
  The CAPS-5 is a clinician-rated PTSD rating scale consisting of 30 items; 20 of these items assess the 20 DSM-5 PTSD symptoms. Symptom cluster scores are calculated as the sum of the individual item severity scores for symptoms contained in a given DSM-5 cluster. These symptom items are scored on a 5-point scale from 0 (absent) to 4 (extreme/incapacitating). Cluster score ranges vary by symptom cluster. Higher scores indicate more severe PTSD symptoms. Therefore, a decrease in the cluster score indicates symptom improvement.
Change from baseline in the PTSD Checklist for DSM-5 (PCL-5) at Day 29, Day 15, and all other timepoints | 8 days, 15 days, 22 days, 29 days, 35 days, and 43 days
  The PCL-5 is a patient-reported PTSD rating scale consisting of 20 items; these items assess the 20 DSM-5 PTSD symptoms. These symptom items are scored on a 5-point scale from 0 (not at all) to 4 (extremely). The total score of the 20 items ranges from 0 to 80 with higher scores indicating more severe PTSD symptoms. Therefore, a decrease in the total score indicates symptom improvement.
Change from baseline in the Sheehan Disability Scale (SDS) at Day 29, Day 15, and Day 43 | 15 days, 29 days, 43 days
  The SDS is a patient-reported measure of disability. The SDS is a composite of 3 items designed to measure the extent to which 3 major domains in the patient's life are functionally impaired by psychiatric or medical symptoms: work, social life/leisure activities, and family life/home responsibilities. Each domain is rated on an 11-point scale from 0 (not at all) to 10 (extremely). The total score is calculated as the sum of the domain scores and ranges from 0 to 30. Higher scores indicate greater disability. Therefore, a decrease in the total score or on individual domains indicates less disability.
Patient Global Impression-Improvement (PGI-I) score at Day 29, Day 15 and all other time points | 8 days, 15 days, 22 days, 29 days, 35 days, and 43 days
  The PGI-I scale is a global self-assessment used to rate the response of a participant's condition to therapy or intervention. It consists of 1 question that asks the participant to rate their current condition compared to how it was prior to beginning treatment on a scale of 1 (very much better) to 7 (very much worse).
Change from baseline in the Insomnia Severity Index (ISI) at Day 29, Day 15, and all other timepoints | 8 days, 15 days, 22 days, 29 days, 35 days, and 43 days
  The ISI is a patient-reported measure of insomnia consisting of 7 items assessing the nature, severity, and impact of insomnia. These items are scored on a 5-point scale from 0 (no problem) to 4 (very severe problem). The total score ranges from 0 to 28 with higher scores indicating more severe insomnia. Therefore, a decrease in the total score indicates symptom improvement.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Praxis Research Site, Phoenix, Arizona
  - Praxis Research Site, Little Rock, Arkansas
  - Praxis Research Site, Rogers, Arkansas
  - Praxis Research Site, Lemon Grove, California
  - Praxis Research Site, Westlake Village, California
  - Praxis Research Site, Fort Myers, Florida
  - Praxis Research Site, Decatur, Georgia
  - Praxis Research Site, Boston, Massachusetts
  - Praxis Research Site, Las Vegas, Nevada
  - Praxis Research Site, Cincinnati, Ohio
  - Praxis Research Site, Dayton, Ohio
  - Praxis Research Site, Oklahoma City, Oklahoma
  - Praxis Research Site, Allentown, Pennsylvania
  - Praxis Research Site, Media, Pennsylvania
  - Praxis Research Site, Austin, Texas
  - Praxis Research Site, Dallas, Texas
  - Praxis Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No